CLINICAL TRIAL: NCT06912945
Title: Factors Affecting the Outcomes of Using the Diode Laser in Benign Laryngeal Lesions
Brief Title: Factors Affecting Outcomes of Using Diode Laser Both 980 nm Wave Length and 450 Wavelength on Benign Laryngeal Lesions in Comparison to Traditional Cold Instrumentations as Regard Parameters of Laser Device, Nature of Lesion and Patient Factors
Acronym: LASER
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelsamei Abdelgalil, Assistant Lecturer of Otorhinolaryngology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-12-3MD
Record Dates: First submitted 2025-03-25; First posted 2025-04-06 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Benign Laryngeal Lesion
Keywords: diode; benign; laryngeal; laser
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (A) (Active Comparator): using diode laser 980nm wavelength in benign laryngeal lesions
  Interventions: Procedure: using diode laser 980nm wavelength in benign laryngeal lesions
- Group (B) (Active Comparator): using diode laser 450nm wavelength in benign laryngeal lesions
  Interventions: Procedure: using diode laser 450nm wavelength in benign laryngeal lesions
- Group (C) (Active Comparator): using traditional cold instrumentations in benign laryngeal lesions
  Interventions: Procedure: using traditional cold instrumentations in benign laryngeal lesions

INTERVENTIONS:
Procedure: using diode laser 980nm wavelength in benign laryngeal lesions — using diode laser 980nm wavelength in treatment of benign laryngeal lesions
  Arms: Group (A)
Procedure: using diode laser 450nm wavelength in benign laryngeal lesions — using diode laser 450nm wavelength in treatment of benign laryngeal lesions
  Arms: Group (B)
Procedure: using traditional cold instrumentations in benign laryngeal lesions — using traditional cold instrumentations in treatment of benign laryngeal lesions
  Arms: Group (C)

SUMMARY:
Studying the different Factors affecting the outcomes of using diode laser both 980 nm wave length and 450 wavelength on benign laryngeal lesions in comparison to traditional cold instrumentations

ELIGIBILITY:
Inclusion Criteria:

- All patients with benign laryngeal lesions

Exclusion Criteria:

* patients presenting with or have history of malignant laryngeal lesion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
change in voice handicap index Arabic version (VHI-Arabic) | 2 months after treatment
  change in Voice handicap index Arabic version from baseline before treatment and after treatment
change in voice acoustic analysis | 2 months after treatment
  change in voice acoustic analysis including change in jitter and shimmer values from baseline preoperative and 2 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abdu Elsamea, Assistant lecturer, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arroyo HH, Neri L, Fussuma CY, Imamura R. Diode Laser for Laryngeal Surgery: a Systematic Review. Int Arch Otorhinolaryngol. 2016 Apr;20(2):172-9. doi: 10.1055/s-0036-1579741. Epub 2016 Mar 4. PMID 27096024